CLINICAL TRIAL: NCT00479349
Title: An Ascending Multiple Dose Study of the Safety, Pharmacokinetics (PK), and Pharmacodynamics (PD) of SAM-531 Administered Orally to Healthy Japanese Young Male and Elderly Subjects
Brief Title: Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of SAM-531
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3193A1-1104
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 1 (Active Comparator): SAM 531 + placebo
  Interventions: Drug: SAM-531

INTERVENTIONS:
Drug: SAM-531 — Multiple ascending doses of SAM 531: 1,5; 3 and 5 mg.

SUMMARY:
To assess the safety and tolerability of ascending multiple oral doses of SAM-531, an investigational drug, in healthy Japanese young male and elderly subjects.To provide the pharmacokinetics (PK) and pharmacodynamics (PD) profiles of multiple oral doses of SAM-531 in healthy Japanese young male and elderly subjects.

ELIGIBILITY:
Inclusion criteria

* Men aged 20 to 45 years, inclusive, at screening.
* Elderly men or women aged 65 years and above as of screening.
* Body mass index (BMI) in the range of 17.6 to 26.4 kg/m2 and body weight ≥45 kg.

Exclusion critereia

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Any clinically important deviation from normal limits in physical examination, vital signs, 12-lead ECGs, or clinical laboratory test results. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels should be below the upper limit of normal at screening.
* Tobacco use or consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or carbonated beverages) or alcoholic beverages within 48 hours before study day 1 until the end of the inpatient confinement period.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 9 months

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tokyo, Japan